CLINICAL TRIAL: NCT02435693
Title: Evaluation of Pharmaceutical Care Program for Type 2 Diabetes Mellitus in Dhule
Brief Title: Pharmaceutical Care Program for Type 2 Diabetes Mellitus
Acronym: pcp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TABREJ MUJAWAR (Other)
Responsible Party: Sponsor-Investigator, TABREJ MUJAWAR, tabrej mujawar mpharm Study principal investigator, R. C. Patel Institute of Pharmaceutical Education & Research
Organization: R. C. Patel Institute of Pharmaceutical Education & Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: pc
Record Dates: First submitted 2015-02-07; First posted 2015-05-06 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: DIABETES MELLITUS, TYPE 2
Keywords: pharmaceutical care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PHARMACEUTICAL CARE programe (Experimental): The pharmaceutical care program was characterized by face to face monthly visits to collect information, register information, prepare plan of care for every health problem; identification of drug therapy problems, communication to prescribers the drug therapy problems identified and education of participants to resolve the drug therapy problems.
  Interventions: Other: PHARMACEUTICAL CARE programe
- control (Other): without pharmaceutical care programe (control)
  Interventions: Other: Without PHARMACEUTICAL CARE programe

INTERVENTIONS:
Other: PHARMACEUTICAL CARE programe — The pharmaceutical care program was characterized by face to face monthly visits to collect information, register information, prepare plan of care for every health problem; identification of drug therapy problems, communication to prescribers the drug therapy problems identified and education of participants to resolve the drug therapy problems.
  Arms: PHARMACEUTICAL CARE programe
Other: Without PHARMACEUTICAL CARE programe
  Arms: control

SUMMARY:
Evaluation of Pharmaceutical Care Program for Type 2 diabetes mellitus in Dhule

Objectives:-

1. To evaluate Pharmaceutical care program in Type2 diabetics.
2. To evaluate the impacts of Pharmaceutical care on quality of life (QOL) in patient with Type-2 Diabetes Mellitus.
3. To study the prevalence of Type2 diabetics cases in Dhule.
4. To study the Assessment of different type of adverse drug reactions (ADRs). In Type2 diabetics.
5. To evaluate the Drug Drug intereaction in Type-2 Diabetes Mellitus.
6. To study the impacts of Pharmaceutical care program on glycemic control in patients with Type-2 Diabetes Mellitus.
7. To study the Drug utilization pattern in Type-2 Diabetes Mellitus in civil hospital Dhule.
8. To compare the efficiency of Pharmaceutical care program and drug in patients with Type-2 Diabetes Mellitus.
9. To study the Pharmaco-economic evaluation in Type-2 Diabetes Mellitus patient's.
10. To increase the patient compliance and positive attitude of patients towards the diabetes disease by counseling.

DETAILED DESCRIPTION:
To evaluate the impacts of Pharmaceutical care on quality of life (QOL) in patient with Type-2 Diabetes Mellitus.

To study the prevalence of Type2 diabetics cases in Dhule. To study the Assessment of different type of adverse drug reactions (ADRs). In Type2 diabetics.

To evaluate the Drug Drug intereaction in Type-2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Patients with type 2 diabetes mellitus of either
* Patients with HbA1c more than 7% and
* Patients with blood sugar level more than 140 mg / dl

Exclusion Criteria:

* Patient with end stage kidney disease.
* Patient with heart failure.
* Patient with chronic Diabetes problem and orthopedic problem

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose measurements recorded (mg/dl).Postprandial blood glucose Recorded: Fasting blood glucose measurements recorded (mg/dl).Postprandial bloodglucoseRecorded | 24 weeks
  Fasting blood glucose measurements recorded (mg/dl).Postprandial blood glucose Recorded Fasting blood glucose measurements recorded (mg/dl).Postprandial blood glucose Recorded fasting blood glucose

SECONDARY OUTCOMES:
Quality of Life score | 24 weeks
  Quality of Life score

CONTACTS AND LOCATIONS:
Overall Officials: tabrej aj mujawar, mpharm, Principal Investigator — muhs
Locations (1):
- Tabrej Aj Mujawar, Dhule, Maharashtra, India